CLINICAL TRIAL: NCT05721950
Title: A Real-World Study to Evaluate the Effectiveness and Safety of Brigatinib in First Line in Patients With ALK Positive Locally Advanced or Metastatic NSCLC in China: An Ambispective, Non-interventional, Observational, Multi-center Study.
Brief Title: A Study to Learn About Brigatinib Treatment Information Available in Chinese Participants With Non-Small-cell Lung Cancer (NSCLC)
Acronym: Brilliant
Status: Active, not recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Brigatinib-4002
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: Drug Therapy; Real-world Data; Anaplastic Lymphoma Kinase Tyrosine Kinase Inhibitors
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — brigatinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Biospecimens collected would be blood and urine samples. They would be used for blood biochemistry coagulation function tests, ALK genetic testing methods and results, and post-resistance gene testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Brigatinib 90 mg/180mg: Participants with ALK positive locally advanced or metastatic NSCLC will be observed ambispectively (retrospective plus prospective) after receiving recommended dose of brigatinib, 90 mg orally once daily for first 7 days followed by 180 mg once daily for up to 36 months as their first line of treatment as part of routine medical care. Data will be collected every 3 months after their first dose until the 36 month or participant death, loss to follow-up, or withdrawal from the study for any reason in the real-world setting from September 1, 2022.
  Interventions: Drug: Brigatinib

INTERVENTIONS:
Drug: Brigatinib — Brigatinib Tablets
  Other Names: Alunbrig

SUMMARY:
The main aim of this study is to learn about the time between the start and stop of treatment with brigatinib in Chinese participants with non-small-cell lung cancer (NSCLC) and who have been positively diagnosed with having the anaplastic lymphoma kinase (ALK) gene. Other study aims are to learn about the progression of NSCLC and participants' response to treatment with brigatinib.

DETAILED DESCRIPTION:
This is a non-interventional, ambispective (retrospective + prospective) study of Chinese participants with ALK-positive locally advanced or metastatic NSCLC receiving brigatinib as their first line of treatment from September 1, 2022.This study will evaluate the time-to-treatment discontinuation and other efficacy outcomes of brigatinib in participants with NSCLC in real-world settings.

This study will enroll approximately 200 participants in the following cohort:

• Brigatinib 90 mg/180mg

This study is an ambispective study that will have prospective data collection if participants enrolled after the study initiation or it will have retrospective data collection if the participants have already started receiving brigatinib as first line treatment before study initiation.

This multi-center trial will be conducted in China. Participants will be followed up for safety from signing informed consent until 36 months after the last dose of treatment or until death of the last participant. The overall time for data collection is approximately 8 years.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 18 years.
2. Participant with histologically/cytologically confirmed locally advanced or metastatic NSCLC.
3. Participants with ALK gene rearrangement confirmed by local hospital medical records.
4. Participants who received brigatinib since September 1, 2022 as first line treatment confirmed by medical records.
5. Participants who have at least one medical record after the start of brigatinib treatment.

Exclusion Criteria

1. Participants participated in NSCLC-related interventional clinical trials after locally advanced or metastatic NSCLC diagnosis and during brigatinib treatment.
2. Previously received any other TKIs, including ALK-targeted TKIs.
3. Previously received more than 1 regimen of systemic anticancer therapy for locally advanced or metastatic disease.
4. Participants have been diagnosed as malignancies (excluding completely resected basal cell carcinoma, bladder carcinoma in situ, cervical carcinoma in situ) in addition to NSCLC within the past 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with ALK positive locally advanced or metastatic NSCLC who received/will receive brigatinib in first line treatment since September 1, 2022 in China.
Sampling Method: Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2024-01-17 (Actual); Primary Completion 2028-03-20 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Real-World Time-to-Treatment Discontinuation (rwTDD) | Up to 8 years
  rwTTD is defined as the time from initiation of brigatinib to discontinuation of treatment for any reason, including disease progression, death, serious adverse events, or participant preference.

SECONDARY OUTCOMES:
Real-World Progression-Free Survival (rwPFS) | Up to 8 years
  rwPFS is defined as the time from initiation of brigatinib to disease progression or death from any cause, or the time of the last confirmed survival.
Real-World Progression-Free Survival at Years 1, 2 and 3 | Up to 8 years
  rwPFS at years 1,2 and 3 is defined as the probability of progression-free survival/ survival over one year; the probability of progression-free survival/survival over two years; the probability of progression-free survival/survival over three years.
Real-World Overall Survival (rwOS) at Years 1, 2 and 3 | Up to 8 years
  rwOS is defined as the time from initiation of brigatinib to death from any cause, or the time of the last confirmed survival.
Real-World Objective Response Rate (rwORR) | Up to 8 years
  rwORR is defined as the percentage of participants who are confirmed to achieved complete response (CR) or partial response (PR) after receiving brigatinib.
Real-World Duration of Response (rwDOR) | Up to 8 years
  rwDOR is defined as the time from the first assessment of CR or PR after receiving first line treatment with brigatinib to progression or death.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Department of Oncology, Shanghai pulmonary hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language. — https://clinicaltrials.takeda.com/study-detail/a4a0ed12fe314db1?idFilter=%5B%22Brigatinib-4002%22%5D